CLINICAL TRIAL: NCT02826278
Title: Study Protocol: Reference Values for External Genitalia and Androgen Blood Level in New Born Girls
Brief Title: Genitalia and Androgen in New Born Girls
Acronym: VOGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL14_0451
Record Dates: First submitted 2016-07-05; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Newborn Genitalia
Keywords: Newborn genitalia; reference charts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy female newborns: Healthy female newborns 24 to 41 weeks of pregnancy without sexual development disturbances
  Interventions: Other: External genitalia measurements in female newborns

INTERVENTIONS:
Other: External genitalia measurements in female newborns

SUMMARY:
Normal values for female external genitalia size at birth, particularly clitoris and blood level of androgens are not well known. This study's aim is to collect normal values in 180 newborn girls of 24 to 41 weeks of pregnancy, and to build genitalia growth charts according to gestational age and birth weight.

The investigators will measure clitoris, genito-anal ratio using a small plastic caliper, at birth, and their evolution until Day 3 of life (if the child is still at the hospital).

The investigators also want to establish normal values of blood testosterone, 17-hydroxyprogesterone, delta4-androstenedione, 21-deoxycortisol, 11-deoxycortisol, deoxycorticosterone, corticosterone, dehydroepiandrostenedione, and dihydrotestosterone), using samples taken for systematic post natal screening of diseases (only in new born of 35 or more weeks of birth).

This is an observational prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female newborns 24 to 41 weeks of pregnancy without sexual development disturbances. Dysmature children - i.e. those with a - 2DS birth weight or height at are not excluded.

Exclusion Criteria:

* Sexual development abnormality, diagnosed pre- or post- birth, endocrine disorder, obstetric trauma affecting genitalia, malformation syndrome, midline abnormalities, congenital cancer, maternal ovary or adrenal tumor diagnosed during pregnancy, mother or father's treatment during pregnancy likely to virilize the fetus, family history of congenital adrenal hyperplasia or neurofibromatosis

Max Age: 3 Days | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Female newborns, with gestational ages of 24 to 41 weeks of pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
length of the clitoris | Day 1
  The measurement is performed on the supine child, with flexed hips and knees retained by the nurse or the nursery nurse. The clitoris will be delimited using cavernosa palpation. The clitoris length will be measured from maxima lablias'root to the top of clitoris, excluding cutaneous cover. Measurements are performed using an-8 cm plastic caliper.
length of the clitoris | Day 3
  The measurement is performed on the supine child, with flexed hips and knees retained by the nurse or the nursery nurse. The clitoris will be delimited using cavernosa palpation. The clitoris length will be measured from maxima lablias'root to the top of clitoris, excluding cutaneous cover. Measurements are performed using an-8 cm plastic caliper

SECONDARY OUTCOMES:
clitoris width | Day 1
  The clitoris will be measured at its base, using an-8 cm plastic caliper.
clitoris width | Day 3
  Measurement will be done if newborns stay at the hospital
anogenital ratio | Day 1
  The ano-genital ratio is the ratio between 1) the distance from anus center to the base of clitoris and 2) the distance from anus center and the posterior commissure of the vulva frenulum.
anogenital ratio | Day 3
  Measurement will be done if newborns stay at the hospital
Blood level of testosterone | Day 3
  This dosage will be performed using a 1.5 ml blood sample taken for screening purpose (for routine systematic post natal screening) only in newborn over 35 WA
Blood level of 17-hydroxyprogesterone | Day 3
  This dosage will be performed using a 1.5 ml blood sample taken for screening purpose (for routine systematic post natal screening) only in newborn over 35 WA
Blood level of delta4-androstenedione | Day 3
  This dosage will be performed using a 1.5 ml blood sample taken for screening purpose (for routine systematic post natal screening) only in newborn over 35 WA
Blood level of 21-deoxycortisol | Day 3
  This dosage will be performed using a 1.5 ml blood sample taken for screening purpose (for routine systematic post natal screening) only in newborn over 35 WA
Blood level of corticosterone | Day 3
  This dosage will be performed using a 1.5 ml blood sample taken for screening purpose (for routine systematic post natal screening) only in newborn over 35 WA
Blood level of dihydrotestosterone | Day 3
  This dosage will be performed using a 1.5 ml blood sample taken for screening purpose (for routine systematic post natal screening) only in newborn over 35 WA

CONTACTS AND LOCATIONS:
Overall Officials: Claire-Lise GAY, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopital Femme Mere Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No